CLINICAL TRIAL: NCT06803498
Title: Delivery Room Intervention and Evaluation (DRIVE) Network
Brief Title: Delivery Room Intervention and Evaluation Network
Acronym: DRIVE Network
Status: Recruiting | Type: Observational
Sponsor: American Academy of Pediatrics (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 21 FO 01
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Resuscitation; Infant, Newborn
Keywords: Continuous Positive Airway Pressure; Intermittent Positive Pressure Ventilation; Intubation, Intratracheal; Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- DRIVE Network Cohort: All infants who receive significant resuscitation intervention (CPAP, PPV, intubation, or CPR) at birth in a DRIVE Network member hospital.
  Interventions: Procedure: Receipt of significant resuscitation intervention at birth

INTERVENTIONS:
Procedure: Receipt of significant resuscitation intervention at birth — Receipt of CPAP, PPV, intubation, or CPR at birth in a hospital delivery room

SUMMARY:
The American Academy of Pediatrics (AAP) convened the multi-center Delivery Room Intervention and Evaluation (DRIVE) Network to establish essential infrastructure to collect, coordinate, and analyze core demographic, resuscitative, and outcome data for an inclusive and diverse population of infants who receive delivery room resuscitation at participating centers. The DRIVE Network consists of delivery hospitals across the United States, covering a range of geographic, urban/rural, racial/ethnic diversity across the country. Together, DRIVE seeks to compare practice-level delivery system characteristics, identify best practices, evaluate outcomes from various interventions, and promote professional development through dissemination via the wide reach of the Neonatal Resuscitation Program.

DETAILED DESCRIPTION:
Basic neonatal resuscitation, which includes drying, warmth, stimulation, suctioning of the baby's nose/mouth as needed, and PPV, comprise the essential skills to which 95% of babies will respond and breathe, yet more data are collected about advanced resuscitative measures that occur in only 3-5% of deliveries. Existing neonatal networks and registries focus on high-risk and premature infants and are not all-inclusive of newborn babies and the basic neonatal resuscitation interventions which save the most lives, but about which little data have been collected in a standardized way. Studying quality of care at birth is also important as it is well known that there is variation between centers, as well as long-standing disparities in infant mortality in the United States.

The objective of this project is to establish essential infrastructure to collect and coordinate core demographic, resuscitative, and outcome variables in an inclusive and diverse population of infants at participating centers. The overarching goal is to relay data back to individual centers, benchmarking their own results against the entire network. Individual centers can employ quality improvement techniques to target professional development activities and improve resuscitation practices. AAP would also use these data to continually improve the educational framework around NRP. Additionally, external investigators could also submit proposals to query the network database on important research questions involving neonatal resuscitation.

ELIGIBILITY:
Inclusion Criteria:

Inborn infant in receipt of a significant resuscitation intervention (CPAP, PPV, intubation, or CPR) at birth

Exclusion Criteria:

Not live born

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All inborn infants who receive significant intervention (CPAP, PPV, intubation, or CPR) at birth in a DRIVE member hospital are included in the DRIVE Database. In addition, summary data is also collected on monthly delivery volume at all sites (stratified by gestational age) to allow for more precise incidence estimates of resuscitative interventions.
Sampling Method: Non-Probability Sample
Enrollment: 3000000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2042-01-01 (Estimated); Study Completion 2042-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient disposition | Immediately after the resuscitation intervention
  The disposition of the patient after resuscitation including newborn nursery, neonatal ICU including a special care nursery or transitional nursery, palliative care, or transfer to other hospital

SECONDARY OUTCOMES:
In-hospital mortality | Within 30 days after birth
  Whether the patient died following resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Foglia, MD MSCE MA FAAP, Principal Investigator — Perelman School of Medicine at the University of Pennsylvania; Beena Kamath-Rayne, MD MPH FAAP, Principal Investigator — American Academy of Pediatrics
Locations (1):
- American Academy of Pediatrics, Itasca, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
For investigators interested in using DRIVE data for observational research, research proposals will be accepted, reviewed, and approved by the DRIVE Steering Committee. Once appropriate regulatory and data use agreements are in place, fully de-identified analytic datasets will be shared for approved protocols. Additionally, at least one DRIVE Steering Committee member will work with the study investigators as a liaison to support the investigators.
Time Frame: Estimated to start in January 2025